CLINICAL TRIAL: NCT07190092
Title: Deep Anterior Cerebellar Stimulation in Treatment of Poststroke Spasticity and Motor Function Impairment.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jan Biziel University Hospital No 2 in Bydgoszcz (Other)
Responsible Party: Principal Investigator, Pawel Sokal, Head of Department of Neurosurgery and Neurology, Jan Biziel University Hospital No 2 in Bydgoszcz
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KB 314/2023
Record Dates: First submitted 2025-09-01; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Post Stroke Spasticity; Dystonia
Keywords: dentate nucleus; DRTt; dentate-rubro-thalamic tract; deep brain stimulation; post-stroke spasticity; rehabilitation
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-frequency stimulation (Experimental): Patients in this arm of the study will undergo implantation of deep brain stimulation electrodes. The stimulation parameters will include a frequency of 130 Hz, which differentiates this arm from the others. The study duration will be four weeks. At the beginning and end of participation in this arm, patients will be examined and assessed using the previously discussed scales.
  Interventions: Procedure: Deep brain stimulation electrode implantation with an electrode target in the dentate nucleus
- Low-frequency stimulation (Experimental): Patients in this arm of the study will have deep brain stimulation electrodes implanted. Stimulation parameters will include a frequency of 50 Hz, which differentiates this arm from the others. The study duration will be four weeks. At the beginning and end of participation in this arm, patients will be examined and assessed using the previously discussed scales.
  Interventions: Procedure: Deep brain stimulation electrode implantation with an electrode target in the dentate nucleus
- No stimulation (Sham Comparator): Patients participating in this arm of the study will have deep brain stimulation electrodes implanted. The stimulation will be turned off. The study will last four weeks. At the beginning and end of their participation in this arm, patients will be assessed and rated using the scales discussed earlier.
  Interventions: Procedure: Deep brain stimulation electrode implantation with an electrode target in the dentate nucleus

INTERVENTIONS:
Procedure: Deep brain stimulation electrode implantation with an electrode target in the dentate nucleus — The intervention will involve implantation of a directional electrode with a target in the dentate nucleus of the cerebellum, ipsilateral to the limbs affected by spasticity. Electrode implantation will be performed using a stereotaxic frame, following prior planning of the electrode trajectory and tractography of the dento-ruborothalamic tract using a planning station. The procedure will be performed under general anesthesia. The IPG stimulator will be placed in the subclavicular region.

SUMMARY:
The aim of this clinical trial is to determine whether deep brain stimulation (DBS) interventions improve rehabilitation and functional recovery in patients with post-stroke spasticity who meet the other inclusion criteria listed below.

Primary question(s) to be answered:

Is DBS stimulation effective in treating post-stroke spasticity? What stimulation frequency is most effective in treating post-stroke spasticity?

Study participants will:

* Undergo surgery to implant a DBS electrode targeting the DRTt (dentate-rubro-thalamic tract ) in close proximity of the dentate nucleus of the cerebellum ipsilateral to the spastic side of the body.
* Each patient will then receive an initial stimulation frequency of 130 Hz (arm 1) and will be assigned to a 4- to 6-week rehabilitation program. After this period, the participant will return for a follow-up visit for a clinical evaluation.
* The frequency will then be changed to 70Hz (arm 2). Patients who have undergone this change will also undergo a rehabilitation period of 4 to 6 weeks. After this period, they will return to the Clinic for a follow-up evaluation.
* The frequency will then be changed to 30Hz (arm 3). Patients who have undergone this change will also undergo a rehabilitation period of 4 to 6 weeks.

Researchers will compare the results obtained from patients in each arm to determine the clinical effects of stimulation and whether they are dependent on the stimulation frequency.

ELIGIBILITY:
Inclusion Criteria:

* One time stroke that occurred 9-36 months ago
* Ischemic or hemorrhagic stroke
* Spastic paresis of at least one limb
* At least 3 months of poststroke rehabilitation in the past
* No improvement of spasticity/motor function for at least 3 months

Exclusion Criteria:

* Seizures after the stroke
* Depression
* Severe sensory deficits
* Anosognosia
* Moderate to severe hemispatial neglect
* Others contraindications for the DBS procedure, e.g. coagulopathy, decompensated chronic disease, etc.
* Contraindication for MRI
* No poststroke rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Increase of FMA score after the rehabilitation with stimulation dentate-rubro-thalamic tract. | 6 weeks
  Increase of FMA score after the rehabilitation

SECONDARY OUTCOMES:
Decrease of Ashworth Scale score after the rehabilitation with dentate-rubro-thalamic tract | 6 weeks
  Decrease of Ashworth Scale score
Improvement in motor function achieves in Motor Assessment Scale MAS with stimulation dentate-rubro-thalamic tract | 6 weeks
  Improvement in motor function achieves in Motor Assessment Scale
Improvement in Modified Rankin Scale after the rehabilitation with stimulation of dentato-rubro-thalamic tract | 6 weeks
  Improvement in Modified Rankin Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery and Neurology University Hospital nr 2 Collegium Medicum Nicolaus Copernicus University, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR